CLINICAL TRIAL: NCT07113418
Title: Role of Fibroblast Growth Factor 21(FGF21) in Breast Cancer
Brief Title: Role of FGF21 in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mostafa Ali, Doctors, Assiut University
Other Study IDs: FGF21 in breast cancer
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients: Female patients admitted at south Egypt cancer institute who diagnosed as breast cancer based on full clinical, radiological and pathological data.
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Enzyme-Linked Immunosorbent Assay. It's a lab technique used to detect and measure specific proteins like antibodies or antigens in a biological sample using enzyme-linked antibodies. When a substrate is added, the enzyme causes a color change, which makes it easy to measure the result accurately.

SUMMARY:
The present study aims to evaluate the serum level of FGF-21 in patients with breast cancer and its correlation with clinical, laboratory, and pathological data.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women, accounting for about 30 %, and its mortality rate is15 % of the incidence rate.

Studies in recent years have shown that the incidence of breast cancer is increasing year by year, which seriously affects Women's quality of life.

Several hormonal. metabolic and inflammatory mechanisms are known to play a role in the development and progression of breast cancer.

Fibroblast growth factor 21 (FGF21) is a protein produced mainly in the liver and regulated by diseases.The elucidation of the endocrine FGF21 signaling pathways in the control of metabolic disease, peroxisome proliferator-activated receptor-α (PPAR-α) which functions in lipid metabolism. However, more data support a versatile role for this molecule acting as a physiologic alert system in several energy homeostasis and their complications has raised great interest and hope in the last year.

Cancer-associated fibroblasts are activated fibroblasts that serve as a key component of the tumor receptors. FGFR1 is often overexpressed in breast and lung cancer, Promoter hypermethylation correlates microenvironment; FGF-19, FGF-21 and FGF-23 are endocrine FGFs that bind to Klotho and FGF with poorer survival of patients.

Clearly, further studies are needed to elucidate the mechanisms behind the increased serum FGF21 levels a high FGF21 secretion by the liver and also by the tumor cells or the stress caused by microenvironment condition that induces an increased FGF21 secretion by mainly the hepatocytes or/and adipocytes in less in cancer patients. It is believed that the elevated FGF21 levels observed in these patients could be due to metabolic disorders. Alternatively, the initiation of the tumor itself could be considered as a stressful degree. A study shows that Circulating FGF-21 level is associated with increased risk of early and late stages of (11)Another study shows that FGF21 is useful as a diagnostic as well as prognostic factor in patients with colorectal carcinogenesis ,supporting a role of inflammation and metabolism atall stages of colorectal carcinogenesis, and suggesting potential use of this biomarker for risk stratification in CRCscreening. endometrioid endometrial carcinoma.

The role of FGF21 in breast cancer and its level is not adequatelyincluded however a study byRanuncolo etal., revealed increased serum level as well astissue expression level of FGF21 in breast cancer.

ELIGIBILITY:
Inclusion Criteria:Female patients admitted at south Egypt cancer institute who diagnosed as breast cancer basedon full clinical, radiological and pathological assays.

-

Exclusion Criteria:Patients diagnosed with other concomitant cancers.

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Female patients admitted at south Egypt cancer institute who diagnosed as breast cancer basedon full clinical, radiological and pathological assays. b. Exclusion criteria:
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Serum FGF21 level measured by ELISA in breast cancer patients compared to healthy controls at enrollment. | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university ( South Egypt Cancer Institute ), Asyut, Egypt

REFERENCES:
- [Background] Gliniak CM, Gordillo R, Youm YH, Lin Q, Crewe C, Zhang Z, Field BC, Fujikawa T, Virostek M, Zhao S, Zhu Y, Rosen CJ, Horvath TL, Dixit VD, Scherer PE. FGF21 promotes longevity in diet-induced obesity through metabolic benefits independent of growth suppression. Cell Metab. 2025 Jul 1;37(7):1547-1567.e6. doi: 10.1016/j.cmet.2025.05.011. Epub 2025 Jun 16. PMID 40527315
- [Background] Cymbaluk-Ploska A, Gargulinska P, Chudecka-Glaz A, Kwiatkowski S, Pius-Sadowska E, Machalinski B. The Suitability of FGF21 and FGF23 as New Biomarkers in Endometrial Cancer Patients. Diagnostics (Basel). 2020 Jun 18;10(6):414. doi: 10.3390/diagnostics10060414. PMID 32570721
- [Background] Ferreira Almeida C, Correia-da-Silva G, Teixeira N, Amaral C. Influence of tumor microenvironment on the different breast cancer subtypes and applied therapies. Biochem Pharmacol. 2024 May;223:116178. doi: 10.1016/j.bcp.2024.116178. Epub 2024 Mar 30. PMID 38561089
- [Background] Ewendt F, Feger M, Foller M. Role of Fibroblast Growth Factor 23 (FGF23) and alphaKlotho in Cancer. Front Cell Dev Biol. 2021 Jan 14;8:601006. doi: 10.3389/fcell.2020.601006. eCollection 2020. PMID 33520985
- [Background] Ping Q, Yan R, Cheng X, Wang W, Zhong Y, Hou Z, Shi Y, Wang C, Li R. Cancer-associated fibroblasts: overview, progress, challenges, and directions. Cancer Gene Ther. 2021 Sep;28(9):984-999. doi: 10.1038/s41417-021-00318-4. Epub 2021 Mar 12. PMID 33712707
- [Background] Sanchez-Hurtado LA, Tejeda-Huezo BC, Gomez-Flores SS, Esquivel-Chavez A, Cano-Oviedo AA, Baltazar-Torres JA. Elderly patients in a Mexican intensive care unit: A retrospective analysis. Med Intensiva (Engl Ed). 2018 May;42(4):258-260. doi: 10.1016/j.medin.2017.03.006. Epub 2017 May 12. No abstract available. English, Spanish. PMID 28502645
- [Background] Gong X, Xiong H, Liu S, Liu Y, Yin L, Tu C, Wang H, Zhao Z, Chen W, Mei Z. Qingpeng Ointment Ameliorates Inflammatory Responses and Dysregulation of Itch-Related Molecules for Its Antipruritic Effects in Experimental Allergic Contact Dermatitis. Front Pharmacol. 2019 Apr 9;10:354. doi: 10.3389/fphar.2019.00354. eCollection 2019. PMID 31024317
- [Background] Luo Y, McKeehan WL. Stressed Liver and Muscle Call on Adipocytes with FGF21. Front Endocrinol (Lausanne). 2013 Dec 18;4:194. doi: 10.3389/fendo.2013.00194. PMID 24385972
- [Background] Falk Libby E, Liu J, Li YI, Lewis MJ, Demark-Wahnefried W, Hurst DR. Globular adiponectin enhances invasion in human breast cancer cells. Oncol Lett. 2016 Jan;11(1):633-641. doi: 10.3892/ol.2015.3965. Epub 2015 Nov 24. PMID 26870258
- [Background] Llovet JM, Montal R, Sia D, Finn RS. Molecular therapies and precision medicine for hepatocellular carcinoma. Nat Rev Clin Oncol. 2018 Oct;15(10):599-616. doi: 10.1038/s41571-018-0073-4. PMID 30061739